CLINICAL TRIAL: NCT03754270
Title: Evaluation of Treatment Effect of Cervical Collar in Moderate Obstructive Sleep Apnea
Brief Title: Cervical Collar for Patients With Moderate Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCMOSA-01
Record Dates: First submitted 2018-10-17; First posted 2018-11-27 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Apnea/hypopnea index
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: The study is a randomized, open, parallel-group intervention study. The two treatment groups are:
  A.Patients with moderate OSA are treated with lifestyle advice (n = 50) B. Patients with moderate OSA are treated with CC and lifestyle advice (n = 50).
  Life style advice is quite subjective and it means that the patients are encouraged to stop smoking, to avoid alcohol, to lose weight, to be more physically active and to avoid sleeping on supine position.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle advice (Active Comparator): Patients receive instructions and advice on lifestyle according to current clinical practice.
  Interventions: Other: Advice in lifestyle
- Lifestyle advice and cervical collar (Experimental): Patients receive the same instructions and advice as in Arm "lifestyle advice" and also get a CC and instructions on how to sleep with it.
  Interventions: Device: Cervical collar

INTERVENTIONS:
Other: Advice in lifestyle — Patients with moderate OSA according to a baseline nocturnal respiratory registration (NRR). Patients receive instructions and advice on lifestyle according to current clinical practice. Life style advice is quite subjective and it means that the patients are encouraged to stop smoking, to avoid alcohol, to lose weight, to be more physically active and to avoid sleeping on supine position.Patients fill in questionnaire 1 that includes questions about nocturnal respiratory disturbances, daytime sleepiness, insomnia, use of tobacco and alcohol, comorbidity and medication. After 6+/-2 weeks of treatment, patients fill in Questionnaire 2 which contains the same questions as Questionnaire 1 and also questions about any side effects, evaluation of treatment. In conjunction with visit 2 another NRR will be performed.
  Arms: Lifestyle advice
Device: Cervical collar — Patients with moderate OSA according to a baseline nocturnal respiratory registration (NRR). Patients receive the same instructions and advice as in Arm "lifestyle advice" and also get a CC and instructions on how to sleep with it. CC is marketed for indications of various diseases such as traumatic cervical injury, cervical disc herniation and other neck problems and allows adjustment of the elevation level to achieve sufficient effect, i.e., extending the neck.Patients fill in questionnaire 1 that includes questions about nocturnal respiratory disturbances, daytime sleepiness, insomnia, use of tobacco and alcohol, comorbidity and medication. After 6+/-2 weeks of treatment, patients fill in Questionnaire 2 which contains the same questions as Questionnaire 1 and also questions about any side effects, evaluation of treatment. In conjunction with visit 2 another NRR will be performed.
  Arms: Lifestyle advice and cervical collar

SUMMARY:
This study evaluates treatment effect of Cervical Collar (CC) in moderate obstructive sleep apnea.The investigators believe that stabilization of the neck by using a CC during sleep helps sustain airway patency. This would mean preventing collapse of airways during sleep.

The study is a randomized, open, parallel-group intervention study. The two treatment groups are:

A. Patients with moderate OSA are treated with lifestyle advice (n = 50) B. Patients with moderate OSA are treated with CC and lifestyle advice (n = 50).

DETAILED DESCRIPTION:
Moderate and severe obstructive sleep apnea (OSA) is strongly associated with cardiovascular diseases, diabetes and also with occupational and traffic accidents due to fatigue and daytime sleepiness. Treatment of moderate OSA is usually by a mandibular advancement device (MAD) and in sometimes even Continuous Positive Airway Pressure (CPAP). MAD and CPAP treatment effectiveness is impeded by limited compliance with long term treatment. Knowledge about mechanical barriers in upper respiratory tract has triggered interest in finding a new treatment method that may prevent collapse of airways during sleep. The investigators believe that stabilization of the neck by using a cervical collar (CC) during sleep helps sustain airway patency. This would mean improved oxygen saturation in the blood and a reduction of daytime fatigue in patients with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Moderate obstructive sleep apnea (AHI 15-30)
* BMI <35
* Age 18-75
* Signed Informed Consent

Exclusion Criteria:

* Ongoing or planned pregnancy during intervention
* Whiplash injury or other neck pain
* Rheumatic diseases
* Dementia
* Active alcohol or drug abuse <2 back in time
* Treatment with sleeping pills or other sedatives
* Cannot wear CC for any reason
* Pregnant or lactating women
* Not expected to be able to comply with nighttime breathing registration/treatment due to medical and/or psychological conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-06-16 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Changes in Apnea Hypopnea Index (AHI) measured at baseline and after 6+/- 2 weeks of treatment. | 6+/- 2 weeks of treatment.
  The definition of AHI is the sum of apneas and hypopneas divided by registration/sleep time. Se below description of Apnea and Hypopnea. According to the international classification of sleep disorders, mild Obstructive Sleep Apnae (OSA) is defined as AHI between 5-15, moderate as AHI between 15-30 and severe sleep apnea as AHI > 30.

OTHER OUTCOMES:
Number of apneas | 6+/- 2 weeks of treatment.
  Apnea is defined as a respiratory arrest during sleep which means more than 90% decrease in respiratory airflow lasting more than 10 seconds with preserved respiratory movement in the thoracic or abdominal wall. This variable is recorded by Nocturnal Respiratory Registration (NRR).
Number of hypopneas | 6+/- 2 weeks of treatment.
  Hypopnea is defined as partial respiratory disturbance during sleep which means a more than 50% decrease in nasal air pressure signal from baseline lasting more than 10. This variable is recorded by Nocturnal Respiratory Registration (NRR).
Variation of body position during sleep | 6+/- 2 weeks of treatment.
  Sleeping in the supine position is increased risk factor that contribute to development of OSA. This variable is recorded by Nocturnal Respiratory Registration (NRR).
Mean level of saturation | 6+/- 2 weeks of treatment.
  OSA cause decrease of oxygen saturation in blood. This variable is recorded by pulse oximeter. Normal pulse oximeter readings usually range from 95 to 100 percent.
Oxygen desaturation index (ODI) | 6+/- 2 weeks of treatment.
  A number of desaturations more than 3% from baseline during sleep divided by number of sleeping hours.This variable is recorded by pulse oximeter.
Percentage of sleeping time with oxygen saturation <90% | 6+/- 2 weeks of treatment.
  It is important för assessing the difference between treatment methods. This variable is recorded by pulse oximeter.
Respiratory rate | 6+/- 2 weeks of treatment.
  It is important for assessing the difference between treatment methods. This variable is recorded by NRR.
Mean heart rate | 6+/- 2 weeks of treatment.
  It is important for assessing the difference between treatment methods. This variable is recorded by NRR.
Quality of life is recorded with 36-item Short Form Health Survey (SF36) | 6+/- 2 weeks of treatment.
  Short Form Health Survey (SF36) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scoring is a two-step process. First, precoded numeric values are recorded per the scoring key given in Table 1. All items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Table 2 lists the items averaged together to create each scale. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Quality of sleep is recorded with adapted questions from Basic Nordic Sleep Questionnaire (BNSQ) | 6+/- 2 weeks of treatment.
  Basic Nordic Sleep Questionnaire (BNSQ) consists of 27 items in 21 different questions and queries a wide range of sleep complaints, including difficulties initiating and maintaining sleep, subjective sleep quality, the use of medication to induce sleep, excessive daytime sleepiness, napping, snoring, and general sleep habits.Sleepiness scores range from 4 to 20 points, insomnia scores from 7 to 35, the higher scores indicating more problems with sleepiness or insomnia.
Sleepiness is recorded with Epworth Sleepiness Scale (ESS) | 6+/- 2 weeks of treatment.
  Epworth Sleepiness Scale (ESS) measures a respondent's general level of daytime sleepiness, or their average sleep propensity in daily life.It is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life.
Tolerability of treatment with CC | 6+/- 2 weeks of treatment.
  It is important for assessing the patient's perception of treatment with CC. This variable is only recorded in experimental arm. There are three simple questions that respondent's should answer:
  "How do you experience treatment in general?" (range very good - very bad), "Do you want to continue with the treatment?" ( yes or no) and "Own comments about the treatment".

CONTACTS AND LOCATIONS:
Overall Officials: Florim Delijaj, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Result] Wang X, Ouyang Y, Wang Z, Zhao G, Liu L, Bi Y. Obstructive sleep apnea and risk of cardiovascular disease and all-cause mortality: a meta-analysis of prospective cohort studies. Int J Cardiol. 2013 Nov 5;169(3):207-14. doi: 10.1016/j.ijcard.2013.08.088. Epub 2013 Sep 8. PMID 24161531
- [Result] Lindberg E, Carter N, Gislason T, Janson C. Role of snoring and daytime sleepiness in occupational accidents. Am J Respir Crit Care Med. 2001 Dec 1;164(11):2031-5. doi: 10.1164/ajrccm.164.11.2102028. PMID 11739131
- [Result] Valham F, Stegmayr B, Eriksson M, Hagg E, Lindberg E, Franklin KA. Snoring and witnessed sleep apnea is related to diabetes mellitus in women. Sleep Med. 2009 Jan;10(1):112-7. doi: 10.1016/j.sleep.2007.11.005. Epub 2008 Jan 22. PMID 18207451
- [Result] Bloom JW, Kaltenborn WT, Quan SF. Risk factors in a general population for snoring. Importance of cigarette smoking and obesity. Chest. 1988 Apr;93(4):678-83. doi: 10.1378/chest.93.4.678. PMID 3258226
- [Result] Farronato G, Storti E, Cuzzocrea ML, Lucchese A, Cossellu G, Assandri F, Biagi R. Three-dimensional changes of the upper airway in patients with obstructive sleep apnea syndrome after a non-adjustable oral appliance treatment. Minerva Stomatol. 2013 Apr;62(4):107-16. English, Italian. PMID 23588211
- [Result] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920
- [Result] Rose EC, Barthlen GM, Staats R, Jonas IE. Therapeutic efficacy of an oral appliance in the treatment of obstructive sleep apnea: a 2-year follow-up. Am J Orthod Dentofacial Orthop. 2002 Mar;121(3):273-9. doi: 10.1067/mod.2002.121006. PMID 11941341
- [Result] Richard W, Venker J, den Herder C, Kox D, van den Berg B, Laman M, van Tinteren H, de Vries N. Acceptance and long-term compliance of nCPAP in obstructive sleep apnea. Eur Arch Otorhinolaryngol. 2007 Sep;264(9):1081-6. doi: 10.1007/s00405-007-0311-3. Epub 2007 Apr 19. PMID 17443336
- [Result] Esclamado RM, Glenn MG, McCulloch TM, Cummings CW. Perioperative complications and risk factors in the surgical treatment of obstructive sleep apnea syndrome. Laryngoscope. 1989 Nov;99(11):1125-9. doi: 10.1288/00005537-198911000-00004. PMID 2530406